CLINICAL TRIAL: NCT01880736
Title: A Trial Investigating the Efficacy and Safety of Flexible vs. Fixed Dosing and Simple vs. Stepwise Titration With Once Daily Insulin Degludec in Inadequately Treated Subjects With Type 2 Diabetes
Brief Title: A Trial Investigating the Efficacy and Safety of Flexible vs. Fixed Dosing and Simple vs. Stepwise Titration With Once Daily (OD) Insulin Degludec in Inadequately Treated Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-4060; U1111-1137-0953 (Other: WHO); JapicCTI- 132164 (Other: JAPIC)
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDeg OD Flexible Dose (Experimental)
  Interventions: Drug: insulin degludec
- IDeg OD Fixed Dose (Experimental)
  Interventions: Drug: insulin degludec
- IDeg OD Simple (Experimental)
  Interventions: Drug: insulin degludec
- IDeg OD Stepwise (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Individual dose adjusted once weekly. IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) to be administered under the skin OD with the option to vary time of administration within a window of plus/minus 8 hours. A maximum of 3 pre-trial OADs are allowed during the trial at an unchanged, stable dose level and dosing frequency.
Drug: insulin degludec — Individual dose adjusted once weekly. IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) to be administered under the skin OD at the same time each day. A maximum of 3 pre-trial OADs are allowed during the trial at an unchanged, stable dose level and dosing frequency.
Drug: insulin degludec — Individual dose adjusted once weekly. IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) to be administered subcutaneously (under the skin) OD at the same time each day. A maximum of 3 pre-trial oral anti-diabetic drugs (OADs) are allowed during the trial at an unchanged, stable dose level and dosing frequency.

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to investigate the efficacy and safety of flexible versus fixed dosing and simple versus stepwise titration with OD insulin degludec in inadequately treated subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Current treatment with IGlar (insulin glargine) with or without OADs (oral antidiabetic drug). All antidiabetic treatments should have been on-going for at least 12 weeks prior to randomisation, and doses of OADs should have been stable in this period of time. - Please note that a maximum of 3 OADs are allowed during this trial: metformin, sulphonylurea (SU)/glinides, dipeptidyl peptidase 4 (DPP-IV) inhibitors, alfa-glucosidaseinhibitors or pioglitazone.
* Diagnosis of T2DM (type 2 diabetes mellitus) at the discretion of the investigator for at least 26 weeks prior to visit 1 (Screening visit)
* HbA1c 7.0-9.5% (both inclusive) by central laboratory analysis
* Body mass index (BMI) equal to or below 35 kg/m^2

Exclusion Criteria:

* Any chronic disorder or severe disease which, in the opinion of the Investigator might jeopardise subject's safety or compliance with the protocol
* Stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty; all within the last 26 weeks prior to Visit 1 (Screening visit)
* Impaired renal function, defined as serum-creatinine higher than or equal to 1.4 mg/dL for males and higher than or equal to 1.3 mg/dL for females
* Current or past (within the last 5 years) malignant neoplasms (except basal cell and squamous cell skin carcinoma)
* Treatment with glucose-lowering agent(s) other than stated in the inclusion criteria in a period of 12 weeks prior to randomisation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (31):
- Japan (31):
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Fukui-shi, Fukui
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Gifu-shi, Gifu
  - Novo Nordisk Investigational Site, Izumisano
  - Novo Nordisk Investigational Site, Kagoshima-shi, Kagoshima
  - Novo Nordisk Investigational Site, Kamakura-shi
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Katsushika-ku, Tokyo
  - Novo Nordisk Investigational Site, Kawasaki-shi, Kanagawa
  - Novo Nordisk Investigational Site, Kitakyushu-shi, Fukuoka
  - Novo Nordisk Investigational Site, Kitakyusyu-shi, Fukuoka
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Niigata-shi, Niigata
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hyogo
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sakaide-shi, Kagawa
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sendai
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yokkaichi-shi, Mie

REFERENCES:
- [Result] Kadowaki T, Jinnouchi H, Kaku K, Herslov ML, Hyllested-Winge J, Nakamura S. Insulin degludec in a simple or stepwise titration algorithm in a Japanese population of patients with type 2 diabetes: a randomized, 26-week, treat-to-target trial. Diabetol Int. 2016 Sep 2;8(1):87-94. doi: 10.1007/s13340-016-0284-9. eCollection 2017 Mar. PMID 30603311
- [Result] Kadowaki T, Jinnouchi H, Kaku K, Herslov ML, Hyllested-Winge J, Nakamura S. Efficacy and safety of once-daily insulin degludec dosed flexibly at convenient times vs fixed dosing at the same time each day in a Japanese cohort with type 2 diabetes: A randomized, 26-week, treat-to-target trial. J Diabetes Investig. 2016 Sep;7(5):711-7. doi: 10.1111/jdi.12502. Epub 2016 Apr 1. PMID 27182031
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 39 sites in Japan.
Pre-assignment Details: Pre-assignment: Subjects switched from their pre-trial IGlar to IDeg unit-to-unit and continued pre-trial OADs (maximum of 3) at unchanged doses and frequency.
Groups:
- IDeg OD Fixed Dosing and Simple Titration (Arm A): The subjects received IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) OD subcutaneously, under the skin of the thigh, upper arm or abdomen for 26 weeks at the same time each day according to the fixed dosing regimen and the simple titration algorithm.
- IDeg OD Fixed Dosing and Stepwise Titration (Arm B): The subjects received IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) OD subcutaneously, under the skin of the thigh, upper arm or abdomen for 26 weeks at the same time each day according to the fixed dosing regimen and the stepwise titration algorithm.
- IDeg OD Flexible Dosing and Simple Titration (Arm C): The subjects received IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) once daily (OD) subcutaneously, under the skin of the thigh, upper arm or abdomen for 26 weeks with the option to vary time of administration within a window of plus/minus 8 hours according to the flexible dosing regimen and the simple titration algorithm.
- IDeg OD Flexible Dosing and Stepwise Titration (Arm D): The subjects received IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) once daily (OD) subcutaneously, under the skin of the thigh, upper arm or abdomen for 26 weeks with the option to vary time of administration within a window of plus/minus 8 hours according to the flexible dosing regimen and the stepwise titration algorithm.
Period: Overall Study
Arm/Group | IDeg OD Fixed Dosing and Simple Titration (Arm A) | IDeg OD Fixed Dosing and Stepwise Titration (Arm B) | IDeg OD Flexible Dosing and Simple Titration (Arm C) | IDeg OD Flexible Dosing and Stepwise Titration (Arm D)
Started | 114 | 115 | 115 | 114
Completed | 113 | 113 | 114 | 108
Not Completed | 1 | 2 | 1 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal Criteria | 1 | 2 | 1 | 5

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects. The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised".
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD Fixed Dosing and Simple Titration (Arm A) | IDeg OD Fixed Dosing and Stepwise Titration (Arm B) | IDeg OD Flexible Dosing and Simple Titration (Arm C) | IDeg OD Flexible Dosing and Stepwise Titration (Arm D) | Total
Number analyzed (Participants) | 114 | 115 | 115 | 114 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.6) | 60.7 (10.5) | 60.0 (10.8) | 60.2 (10.8) | 60.3 (10.7)
Gender [Count of Participants; unit: Participants]
  Female | 41 | 41 | 50 | 34 | 166
  Male | 73 | 74 | 65 | 80 | 292
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.8 (0.6) | 7.8 (0.6) | 7.8 (0.5) | 7.8 (0.6) | 7.8 (0.6)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 129.8 (30.0) | 136.0 (38.1) | 131.8 (33.5) | 134.5 (39.6) | 133.0 (35.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (%) Glycosylated Haemoglobin)
Description: Changes from baseline in HbA1c values over time period of Week 0-26 were evaluated by dosing regimen (flexible vs. fixed dosing) and by titration algorithm (simple vs stepwise)
Time Frame: Week 0, week 26
Population: The full analysis set (FAS) included all randomised subjects. 458 subjects were grouped either according to dosing pattern or treatment algorithm received. Analysis was per intention to treat principle. Missing values were imputed using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Groups:
- IDeg OD Flexible (Arm C+Arm D): The trial followed a 2X2 factorial design and therefore the subjects included in this arm are those who received IDeg in a flexible dosing pattern irrespective of titration algorithm used. The subjects received IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) once daily (OD) subcutaneously, under the skin of the thigh, upper arm or abdomen for 26 weeks with the option to vary time of administration within a window of plus/minus 8 hours according to the flexible dosing regimen. A maximum of 3 pre-trial oral anti-diabetic drugs (OADs) were allowed during the trial at an unchanged, stable dose level and frequency.
- IDeg OD Fixed (Arm A+Arm B): The trial followed a 2X2 factorial design and therefore the subjects included in this arm are those who received IDeg in a fixed dosing pattern irrespective of titration algorithm used. The subjects received IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) OD subcutaneously, under the skin of the thigh, upper arm or abdomen for 26 weeks at the same time each day according to the fixed dosing regimen. A maximum of 3 pre-trial OADs were allowed during the trial at an unchanged, stable dose level and dosing frequency.
- IDeg OD Simple (Arm A+Arm C): The trial followed a 2X2 factorial design and therefore the subjects included in this arm are those who followed simple titration algorithm irrespective of dosing pattern used. The subjects received IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) OD subcutaneously, under the skin of the thigh, upper arm or abdomen for 26 weeks according to the simple titration algorithm. Individual dose was adjusted once weekly was based upon a single pre-breakfast self-measured plasma glucose (SMPG) value measured in the morning of visits 3-27. The dose was either increased by 2 units if pre-breakfast SMPG was above target (4.0-5.0 mmol/L or 71-90 mg/dL) or reduced by 2 units if below target. A maximum of 3 pre-trial OADs were allowed during the trial at an unchanged, stable dose level and dosing frequency.
- IDeg OD Stepwise (Arm B+Arm D): The trial followed a 2X2 factorial design and therefore the subjects included in this arm are those who followed stepwise titration algorithm irrespective of dosing pattern used. The subjects received IDeg (100 U/mL, 3 mL FlexTouch® pen PDS290) OD subcutaneously, under the skin of the thigh, upper arm or abdomen for 26 weeks according to the stepwise titration algorithm. Individual dose was adjusted once weekly and based on the mean of three pre-breakfast SMPG values measured in the morning of titration and the preceding two days. The dose was increased in multiples of 2 units, to a maximum of 8 units, depending on the mean pre-breakfast SMPG value or reduced if symptomatic hypoglycaemia or documented low SMPG values (≤ 3.9 mmol/L/70 mg/dL) occurred. A maximum of 3 pre-trial OADs were allowed during the trial at an unchanged, stable dose level and dosing frequency.
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 229 | 229 | 229 | 229
Percent (%) glycosylated haemoglobin | -0.54 (0.76) | -0.62 (0.75) | -0.57 (0.72) | -0.59 (0.80)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Changes from baseline in FPG values over the time period of Week 0-26 were evaluated by dosing regimen (flexible vs. fixed dosing) and by titration algorithm (simple vs stepwise).
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. 458 subjects were grouped according to dosing pattern or treatment algorithm received. Analysis was per intention to treat principle. Missing values were imputed using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 229 | 229 | 229 | 229
mg/dL | -28.8 (39.0) | -25.4 (40.2) | -27.0 (35.3) | -27.2 (43.6)

3. Secondary Outcome: Responder for HbA1c (%) Based on Central Laboratory Assessment: HbA1c Below 7.0% at End of Trial
Description: The number of subjects who achieved the pre-defined HbA1c target (<7.0%) after 26 weeks of treatment was recorded by dosing regimen (flexible vs. fixed dosing) and by titration algorithm (simple vs stepwise).
Time Frame: After 26 weeks of treatment
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 229 | 229 | 229 | 229
Subjects | 90 | 95 | 91 | 94

4. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: The incidences of treatment emergent adverse events (TEAEs) over the time period of Week 0-26 were recorded by dosing regimen (flexible vs. fixed dosing); and by titration algorithm (simple vs stepwise).
Time Frame: Weeks 0-26
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator. 458 subjects were grouped according to dosing pattern or treatment algorithm received. Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: events
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 229 | 229 | 229 | 229
events | 150 | 154 | 138 | 166

5. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes (Defined as Severe Hypoglycaemia and/or a Measured Plasma Glucose (PG) Less Than 3.1 mmol/L (Less Than 56 mg/dL))
Description: The confirmed hypoglycaemic episodes (defined as severe hypoglycaemia and/or a measured plasma glucose (PG) less than 3.1 mmol/L [less than 56 mg/dL]) over the time period of Week 0-26 was recorded by dosing regimen (flexible vs. fixed dosing); and by titration algorithm (simple vs stepwise).
Time Frame: Weeks 0-26
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator. 458 subjects were grouped either according to dosing pattern or treatment algorithm received. Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: episodes
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 229 | 229 | 229 | 229
episodes | 476 | 371 | 469 | 378

6. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association (ADA) Definition
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA definition (classified as severe hypoglycaemia, documented hypoglycaemia, asymptomatic hypoglycaemia, probable symptomatic hypoglycaemia, relative hypoglycaemia) over the time period of Week 0-26 was recorded by dosing regimen (flexible vs. fixed dosing) and by titration algorithm (simple vs stepwise).
Time Frame: Weeks 0-26
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator. 458 subjects were grouped either according to dosing pattern or treatment algorithm received. Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: episodes
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 229 | 229 | 229 | 229
episodes
  ADA Events Overall | 3053 | 2736 | 3089 | 2700
  Severe | 0 | 1 | 1 | 0
  Documented symptomatic | 1262 | 1141 | 1293 | 1110
  Asymptomatic | 1523 | 1283 | 1505 | 1301
  Probable symptomatic | 87 | 131 | 103 | 115
  Relative | 181 | 180 | 187 | 174

7. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes in the Maintenance Period
Description: The number of treatment mergent confirmed hypoglycaemic episodes in the maintenance period from Week 16 to end of trial (week 27) was recorded by dosing regimen (flexible vs. fixed dosing) and by titration algorithm (simple vs. stepwise). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes with a confirmed plasma glucose value of less than 3.1 mmol/L.
Time Frame: From Week 16 to end of trial (week 27)
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product. Subjects were grouped either according to dosing pattern or treatment algorithm received. 451 subjects contributed to the analysis. Subjects in the safety analysis set contributed to the evaluation "as treated".
Measure: Number; unit: episodes
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 223 | 228 | 227 | 224
episodes | 227 | 192 | 241 | 178

8. Secondary Outcome: Number of Treatment Emergent Nocturnal (00:01-05:59 am) Confirmed Hypoglycaemic Episodes
Description: The number of treatment emergent nocturnal (00:01-05:59 am) confirmed hypoglycaemic episodes over the time period of Week 0-26 was recorded by dosing regimen (flexible vs. fixed dosing) and by titration algorithm (simple vs stepwise). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes with a confirmed plasma glucose value of less than 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Weeks 0-26
Population: as for outcome 6
Measure: Number; unit: episodes
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 229 | 229 | 229 | 229
episodes | 77 | 58 | 80 | 55

9. Secondary Outcome: Number of Treatment Emergent Nocturnal (00:01-05:59 am) Confirmed Hypoglycaemic Episodes in the Maintenance Period
Description: The number of treatment emergent nocturnal (00:01-05:59 am) confirmed hypoglycaemic episodes in the maintenance period from 16 weeks to end of trial (week 27) was recorded by dosing regimen (flexible vs. fixed dosing); and by titration algorithm (simple vs stepwise). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes with a confirmed plasma glucose value of less than 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: From week 16 to end of trial (week 27)
Population: as for outcome 6
Measure: Number; unit: episodes
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Number analyzed (Participants) | 229 | 229 | 229 | 229
episodes | 34 | 23 | 40 | 17

ADVERSE EVENTS:
Time Frame: This included events from the first trial related activity after the subject had signed the informed consent and until the end of the follow-up period (Week 27).
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator. 458 subjects were grouped either according to dosing pattern or treatment algorithm received. Subjects in the safety set contributed to the evaluation "as treated".
Arm/Group | IDeg OD Flexible (Arm C+Arm D) | IDeg OD Fixed (Arm A+Arm B) | IDeg OD Simple (Arm A+Arm C) | IDeg OD Stepwise (Arm B+Arm D)
Serious Adverse Events (participants affected / at risk) | 8/229 | 6/229 | 7/229 | 7/229
Other Adverse Events (participants affected / at risk) | 79/229 | 82/229 | 78/229 | 83/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD Flexible (Arm C+Arm D) (N=229) | IDeg OD Fixed (Arm A+Arm B) (N=229) | IDeg OD Simple (Arm A+Arm C) (N=229) | IDeg OD Stepwise (Arm B+Arm D) (N=229)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD Flexible (Arm C+Arm D) (N=229) | IDeg OD Fixed (Arm A+Arm B) (N=229) | IDeg OD Simple (Arm A+Arm C) (N=229) | IDeg OD Stepwise (Arm B+Arm D) (N=229)
Diabetic retinopathy (Eye disorders) | 24 (25) | 20 (20) | 18 (18) | 26 (27)
Nasopharyngitis (Infections and infestations) | 67 (87) | 69 (92) | 68 (90) | 68 (89)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.